CLINICAL TRIAL: NCT03576547
Title: A Phase I/II Study of the Combination of Venetoclax, Ponatinib and Corticosteroids in Patients With Relapsed or Refractory Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia and Lymphoid Blast Phase Chronic Myelogenous Leukemia
Brief Title: Venetoclax, Ponatinib, and Dexamethasone in Participants With Philadelphia Chromosome or BCR-ABL Positive Relapsed or Refractory Acute Lymphoblastic Leukemia or Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to slow accrual and low level of interest both by the sponsor and by the department
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0313; NCI-2018-01100 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0313 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-26; First posted 2018-07-03 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive; Recurrent Acute Lymphoblastic Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Acute Lymphoblastic Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; t(9;22)
MeSH Terms: conditions — Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ponatinib; Rituximab; CT-P10; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I (400 mg Ponatinib) Treatment (ponatinib, venetoclax, dexamethasone, rituximab) (Experimental): The regimen consists of 4 cycles of induction/consolidation followed by up to 2 years of maintenance therapy for responding patients.
  Interventions: Drug: Dexamethasone; Drug: Ponatinib Hydrochloride; Biological: Rituximab; Drug: Venetoclax
- Phase I (800 mg Ponatinib) Treatment (ponatinib, venetoclax, dexamethasone, rituximab) (Experimental): The regimen consists of 4 cycles of induction/consolidation followed by up to 2 years of maintenance therapy for responding patients.
  Interventions: Drug: Dexamethasone; Drug: Ponatinib Hydrochloride; Biological: Rituximab; Drug: Venetoclax
- Phase II Ponatinib MDT (Experimental): Participants in Phase II will receive the dose that was determined to be the Maximum Tolerated Dose (MDT) found in the Phase I portion of the study. The regimen consists of 4 cycles of induction/consolidation followed by up to 2 years of maintenance therapy for responding patients.
  Interventions: Drug: Dexamethasone; Drug: Ponatinib Hydrochloride; Biological: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ponatinib Hydrochloride — Given PO
  Other Names: AP24534 HCl; Iclusig
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase I/II trial studies the best dose of venetoclax when given together with ponatinib and dexamethasone and to see how well they work in treating participants with Philadelphia chromosome or BCR-ABL positive acute lymphoblastic leukemia or chronic myelogenous leukemia that has come back or does not respond to treatment. Drugs used in chemotherapy, such as venetoclax and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ponatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving venetoclax, ponatinib, and dexamethasone may work better in treating participants with acute lymphoblastic leukemia or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of venetoclax, ponatinib, and dexamethasone in patients with relapsed/refractory Philadelphia positive (Ph+) acute lymphoblastic leukemia (ALL) or lymphoid blastic phase (BP)-chronic myelogenous leukemia (CML). (Phase I) II. To determine the efficacy of the regimen, as defined by the rate of complete remission (CR) or CR with incomplete count recovery (CRi). (Phase II)

SECONDARY OBJECTIVES:

I. To determine efficacy outcomes, including rate of minimal residual disease negativity by polymerase chain reaction (PCR) for BCR-ABL1 transcripts, median relapse-free survival (RFS), and median overall survival (OS).

II. To determine the proportion of patients proceeding to allogeneic stem cell transplant (ASCT).

III. To preliminarily determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To evaluate the effect of single-agent ponatinib on apoptotic proteins and Bcl-2 dependency.

II. To correlate apoptotic protein expression and Bcl-2 dependency on response and resistance to the combination regimen.

III. To assess impact of baseline genomics on outcomes with the combination regimen.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study.

INDUCTION (COURSE 1): Participants who have not received ponatinib within 2 weeks of the anticipated start date receive ponatinib orally (PO) daily on days 1-35, venetoclax PO daily on days 8-35, and dexamethasone PO or intravenously (IV) over 15 minutes on days 8-11. Participants who have received ponatinib within 2 weeks of the anticipated start date receive ponatinib PO and venetoclax PO daily on days 1-28 and dexamethasone PO or IV over 15 minutes on days 1-4. Participants with CD20 expression receive rituximab IV over 2-6 hours on days 14 and 21 at the discretion of the treating physician after the maximum dose of venetoclax has been reached.

CONSOLIDATION (COURSES 2-4): Participants receive ponatinib PO and venetoclax PO daily on days 1-28 and dexamethasone PO or IV over 15 minutes on days 1-4. Participants with CD20 expression receive rituximab IV over 2-6 hours for up to 2 doses each course at the discretion of the treating physician after the maximum dose of venetoclax has been reached. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE (COURSES 5+): Participants receive ponatinib PO and venetoclax PO daily on days 1-28 and dexamethasone PO or IV over 15 minutes on days 1-4. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Participants achieving remission undergo ASCT at the discretion of the treating physician.

After completion of study treatment, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory Ph-positive ALL or lymphoid blast phase CML (either t(9;22) and/or BCR-ABL1 positive by fluorescent in situ hybridization or polymerase chain reaction), including prior therapy with at least one Bcr-Abl tyrosine kinase inhibitor
* Performance status =< 3 Eastern Cooperative Oncology Group (ECOG scale)
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the principal investigator (PI)
* Alanine aminotransferase (ALT) =< 1.5 x ULN, unless due to the underlying leukemia approved by the PI
* Aspartate aminotransferase (AST) =< 1.5 x ULN unless due to the underlying leukemia approved by the PI
* Creatinine clearance >= 30 mL/min
* Serum lipase and amylase =< 1.5 x ULN
* Ability to swallow
* Signed informed consent

Exclusion Criteria:

* Prior history of treatment with venetoclax. Prior ponatinib is allowed
* Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment)
* History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
* Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
* Active secondary malignancy that in the investigator's opinion will shorten survival to less than 1 year
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria
* Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to: any history of myocardial infarction (MI), stroke, revascularization, unstable angina or transient ischemic attack prior to enrollment; left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment; diagnosed or suspected congenital long QT syndrome; any history of clinically significant atrial or ventricular arrhythmias (such as uncontrolled atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) as determined by the treating physician; prolonged corrected QT interval (QTc) interval on pre-entry electrocardiogram (> 480 msec) unless corrected after electrolyte replacement; history of venous thromboembolism including deep venous thrombosis or pulmonary embolism within the past 3 months; uncontrolled hypertension (diastolic blood pressure > 100 mmHg; systolic > 150 mmHg)
* Patients currently taking drugs that are generally accepted to have a high risk of causing Torsades de Pointes (unless these can be changed to acceptable alternatives)
* Received strong or moderate CYP3A inhibitors or inducers within 3 days of study entry
* Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 3 days prior to starting venetoclax
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Prior recent treatment with corticosteroids and hydroxyurea is permitted
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception throughout the study period. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. Appropriate birth control will be determined by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study did not move on from the Phase I portion of this trial. There was no MTD reached and zero participants were registered on Phase II of this study.
Period: Overall Study
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Started | 3 | 6 | 0
Completed | 3 | 6 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study did not move on from the Phase I portion of this trial. There was no MTD reached and zero participants were registered on Phase II of this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT | Total
Number analyzed (Participants) | 3 | 6 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 2 | 3 |  | 5
  >=65 years | 1 | 3 |  | 4
Age, Continuous [Median (Full Range); unit: years] | 35 [26 to 73] | 54 [26 to 71] |  | 37 [26 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 |  | 2
  Male | 2 | 5 |  | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 1 | 1 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 1 |  | 1
  White | 2 | 4 |  | 6
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Venetoclax When Given in Combination With Ponatinib and Dexamethasone (Phase I)
Description: MTD is defined as the highest dose level where a dose limiting toxicity (DLT) occurs within at most one out of six patients treated. The MTD is defined as the highest dose studied for which the observed incidence of DLT is less than 33%. Frequencies of toxicities will be tabulated according to the National Cancer Institute (NCI) Common Toxicity Criteria. Patients will be continued to be followed for one year for evidence of late toxicity.
Time Frame: Up to 1 year
Population: as for baseline characteristics
Measure: Number; unit: Milligrams
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 3 | 6 | 0
Milligrams | NA — Due to insufficient number of participants, the MTD was not reached. | NA — Due to insufficient number of participants, the MTD was not reached. |

2. Primary Outcome: Number of Participants With a Response Complete Response (CR) + CR With Incomplete Count Recovery (CRi)
Description: Overall response rate, defined as the rate or complete response (CR) + CR with incomplete count recovery (CRi). Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR. Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L; neutrophils < 1 x 10^9/L).
Time Frame: 9 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 3 | 6 | 0
Participants | 0 | 5 |

3. Primary Outcome: Event Free Survival (EFS)
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: Monthly up to 5 years, 11 months and 7 days
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 3 | 6 | 0
Months | 1.9 [1.7 to 2.9] | 17.6 [2.7 to 49.1] |

4. Secondary Outcome: Number of Participants Achieving Minimal Residual Disease Negativity
Description: The proportion of patient achieving minimal residual disease negativity (as assessed by polymerase chain reaction PCR for BCR-ABL transcripts) after 2 cycles of therapy will be estimated.
Time Frame: After 2 cycles of therapy
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 3 | 6 | 0
Participants | 0 | 4 |

5. Secondary Outcome: Proportion of Patients Proceeding to Allogeneic Stem Cell Transplant (ASCT) a
Description: All patients assessed for allogeneic stem cell transplant.
Time Frame: Up to 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 3 | 6 | 0
Participants | 0 | 0 |

6. Secondary Outcome: Overall Survival (OS)
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: From treatment initiation to death or last follow-up, up to 5 years, 11 months and 7 days
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 3 | 6 | 0
Months | 5.4 [5.0 to 56.4] | 21.9 [14.4 to 51.6] |

7. Secondary Outcome: Relapse-free Survival (RFS)
Description: Relapse-free survival is the time from documented CR/CRi until relapse or death. Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR. Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L; neutrophils < 1 x 10^9/L).
Time Frame: Monthly up to 5 years, 11 months and 7 days
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
Number analyzed (Participants) | 0 | 5 | 0
Months |  | NA [13.3 to 48.0] — Survival will be presented by median survival, which is the time point at which the cumulative survival drops below 50%. If there is no median survival (not reached), it means the cumulative survival was more than 50%. |

ADVERSE EVENTS:
Time Frame: Up to 5 years, 11 months and 7 days.
Description: This study did not move on from the Phase I portion of this trial. There was no MTD reached and zero participants were registered on Phase II of this study.
Arm/Group | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) | Phase II Ponatinib MDT
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/3 | 6/6 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) (N=3) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) (N=6) | Phase II Ponatinib MDT (N=0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | NA
Fever (General disorders) | 0 (0) | 1 (1) | NA
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | NA
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | NA
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | NA
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | NA
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | NA
Pain (General disorders) | 2 (2) | 0 (0) | NA
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | NA
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (400 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) (N=3) | Phase I (800 mg Ponatinib) Treatment (Ponatinib, Venetoclax, Dexamethasone, Rituximab) (N=6) | Phase II Ponatinib MDT (N=0)
Alanine aminotransferase increased (Investigations) | 2 (6) | 1 (2) | NA
Alkaline phosphatase increased (Investigations) | 2 (6) | 0 (0) | NA
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA
Aspartate aminotransferase increased (Investigations) | 2 (4) | 0 (0) | NA
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | NA
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Eye infection (Eye disorders) | 0 (0) | 1 (1) | NA
Fatigue (General disorders) | 0 (0) | 1 (1) | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | NA
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | NA
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | NA
Neutrophil count decreased (Investigations) | 0 (0) | 4 (7) | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | NA
Platelet count decreased (Investigations) | 0 (0) | 3 (5) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow accrual. The trial did not move on to Phase II, therefore zero participants were registered on the Phase II Portion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03576547/Prot_SAP_001.pdf